CLINICAL TRIAL: NCT02039544
Title: A Randomized, Parallel-controlled, Clinical Study to Evaluate the Efficacy of Xuebi Prescription Compared With Placebo in the Treatment of Diabetic Peripheral Neuropathy(Qi Deficiency and Blood Stasis)
Brief Title: A Study of Xuebi Formula for Diabetic Peripheral Neuropathy(Qi-deficiency and Blood-stasis)
Acronym: XB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Fengmei Lian, chair, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20131205
Record Dates: First submitted 2013-12-08; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetes; Chinese Herbs
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xuebi formula (Experimental): Xuebi formula , one dosage ,every day, treat 6 months.
  Interventions: Drug: Xuebi formula
- Placebo (Placebo Comparator): placebo,has the same taste and color as Xuebi formula one dosage ,every day, treat 6 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Xuebi formula
  Arms: Xuebi formula
Drug: placebo
  Arms: Placebo

SUMMARY:
A Randomized, Parallel-controlled, Clinical Study to Evaluate the Efficacy of Xuebi Prescription Compared With Placebo in the Treatment of Diabetic Peripheral Neuropathy(Qi Deficiency and Blood Stasis)

DETAILED DESCRIPTION:
Charged by the sponsor in line with traditional Chinese medicine Qi deficiency and blood stasis syndrome 60 cases have DPN，they were randomly divided into Chinese herbal compound Xuebi prescription group and placebo group. The treatment groups were compared 24-week composite score.

ELIGIBILITY:
* according to the 1999 WHO criteria, in accordance with the diagnostic criteria for type 2 diabetes.
* according to the diagnostic standard of diabetes peripheral nerve lesions.
* age range 30-70 years.
* Syndrome of traditional Chinese medicine is Qi deficiency and blood stasis.
* FBG < 13.9mmol/L, HbA1c<10%.
* signed the informed consent

Exclusion Criteria:

* did not meet the inclusion criteria, or incomplete information affect the clinical syndrome differentiation type;
* repeated hypoglycemia reaction, nearly a month diabetic ketoacidosis, DKAand severe infections;
* blood pressure without control or after control, SBP ≥ 160mmHg or (and)DBP ≥ 100mmHg;
* TG≥ 5.6mmol / L;
* diabetic lower extremity vascular disease (resting ankle brachial index in patients with ABI ≤ 0.90 or lower extremity ultrasound vascular stenosis > 50%).
* pregnancy, to pregnant or lactating women;
* the ingredients allergy of Chinese herbal medicine and allergic constitution person;
* psychiatric patients;
* have serious heart, lung, liver, kidney, brain and other complications overassociated with other severe primary diseases;
* other patients had participated in clinical trials or are in other clinical trials before the test in January;
* in the past 5 years with alcohol and / or psychoactive substances, drug abuse and dependence;
* according to the researcher's judgment, can reduce the possibility of the group or other diseases or conditions were complicated, such as work environment change frequently, the living environment is not stable, easy to cause lost
* hepatic, renal impairment (ALT, AST is greater than 2.5 times the upper limit of normal value; serum creatinine greater than 1.5 times the upper limit of normal value);
* demyelinating lesions or from other causes of polyneuropathy patients.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change in Scores of TCM clinical symptom and the clinical scoring system of Toronto (TCSS) | 24weeks
  1. Scores of TCM clinical symptom. Using statistical table score, main symptoms and secondary symptoms according to the degree is divided into light, medium, heavy, the main symptoms were recorded 2, 4, 6 points, the secondary symptoms were recorded 1, 2, 3 points. No symptomatic record 0 points. Before the study, of 4, 8, 12, 16, 20, 24 week each recorded 1 times. Description of tongue and pulse only, not scoring.
  2. the clinical scoring system of Toronto (TCSS). TCSS includes a score of neural symptoms, nerve reflex scores and sensory examination , a total of 19 points.Before the study, of 4, 8, 12, 16, 20, 24 week each scoring 1 times.According to the classification standard, 0-5 points does not have DPN, 6-8 points for mild DPN, 9-11 points for moderate DPN, 12-19 points for severe DPN.

SECONDARY OUTCOMES:
Change in Nerve conduction velocity | 24Weeks
  Nerve conduction velocity are recorded at 0,12th,24th weeks.

OTHER OUTCOMES:
Number of participants with adverse events | 24Weeks
  Adverse events with records at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Tong, PHD, Study Chair — Guang'anmen Hospital